CLINICAL TRIAL: NCT06736938
Title: Efficacy and Safety of Balanced Analgosedation in Bronchoscopy With Propofol/Pethidine Versus Midazolam/Pethidine: a Single-centre Randomised Controlled Trial
Brief Title: Balanced Analgosedation in Bronchoscopy: Propofol/Pethidine Versus Midazolam/Pethidine
Acronym: ABroProMida
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Andrea Cesalpino Arezzo ONLUS (Other)
Collaborators: Azienda USL Toscana Sud Est (Other Government); Ospedale San Donato, Arezzo (Unknown)
Responsible Party: Principal Investigator, Raffaele Scala, Head of COU Pulmonology and RICU - San Donato Hospital, Fondazione Andrea Cesalpino Arezzo ONLUS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20245188206500; 2024-518820-65-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-09; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Sedation During Bronchoscopy
Keywords: Balanced Analgosedation; Pulmonologist; Propofol; MIdazolam; Petidhine
MeSH Terms: interventions — Propofol; Midazolam; Meperidine

STUDY DESIGN:
Intervention Model Description: Eligible patients may undergo flexible bronchoscopy based solely on clinical indications, with procedures classified as either interventional (e.g., laser therapy, ndotracheal/endobronchial debulking, visual biopsies, mucosal biopsies, or transbronchial biopsies guided by echo-endoscopy such as EBUS or EUS) or non-bioptic procedures, such as bronchial lavage, bronchoalveolar lavage, or endobronchial lavage. To ensure a balanced distribution of characteristics that could influence study outcomes, stratified block randomisation will be used. Patients will be stratified according to the type of bronchoscopic procedure (interventional vs simple), as the complexity and invasiveness of the procedure may influence the required depth of sedation. Within each group, block randomisation with a 1:1 ratio will be applied to ensure a consistent balance of patients recruited between treatment groups (Propofol+Pethidine or Midazolam+Pethidine).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Bronchoscopy (Active Comparator): eg., laser therapy, endotracheal/endobronchial debulking, visual biopsies, mucosal biopsies, or transbronchial biopsies guided by echo-endoscopy such as EBUS or EUS
  Interventions: Drug: Propofol 1%; Drug: Midazolam; Drug: Pethidine
- Non-bioptic Bronchoscopy (Active Comparator): such as bronchial lavage, bronchoalveolar lavage or endobronchial lavage.
  Interventions: Drug: Propofol 1%; Drug: Midazolam; Drug: Pethidine

INTERVENTIONS:
Drug: Propofol 1% — Propofol 1% is infused intravenously, initially at a bolus dose of 0.5 mg/kg followed by a maintenance dose in a continuous infusion of 0.5-1.0 mg/kg/hour.
Drug: Midazolam — Midazolam is administered intravenously at an initial dose of 2 mg, as a bolus, followed by aliquots of 0.5 mg or 1 mg.
Drug: Pethidine — Pethidine (100 mg/2 ml) is administered intravenously at a dosage of 0.5 mg/kg.

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of two pharmacological sedation regimens during bronchoscopy procedures in adult patients who require elective bronchoscopy.

The main questions it aims to answer are:

* Is propofol/pethidine analgesia administered by a pulmonologist as effective and safe as midazolam/pethidine in achieving adequate sedation during bronchoscopy, particularly in terms of desaturation rate?
* Does the choice of sedative (midazolam vs. propofol) influence the occurrence of adverse events or need for escalated care?

DETAILED DESCRIPTION:
Bronchoscopic procedures are essential in the diagnosis and management of various respiratory diseases, but they can cause significant discomfort for patients.

Analgosedation plays a crucial role in improving patient comfort while ensuring optimal conditions for the safe performance of the procedure. However, sedation management protocols can vary greatly depending on the hospital center and the availability of an anesthetist.

Over the years, with the increasing number of bronchoscopic procedures, the growing complexity of patients-particularly those with pulmonary diseases presenting comorbidities and significant gas exchange alterations-and the limited availability of anesthetists in national hospital facilities, there has been a growing reliance on independently managed procedural sedation.

This independent management-without the need for an anesthesia specialist-has been facilitated by the use of relatively easy-to-manage drugs like midazolam, a benzodiazepine (BDZ) with a pharmacokinetic profile that makes it preferable to other similar compounds due to its rapid onset of action and the availability of an antagonist capable of reversing its effects.

However, it is important to acknowledge that the use of midazolam carries significant risks.

Propofol, compared to midazolam, is characterized by an even faster onset of action, but more importantly by higher clearance and redistribution, allowing for rapid recovery of consciousness even after prolonged infusions. Nevertheless, this drug is also associated with adverse effects, particularly on cardiac inotropic and chronotropic function as well as mean arterial pressure, thus requiring caution in its administration.

The use of propofol-as per the technical data sheet approved by the Italian Medicines Agency (AIFA)-is reserved for doctors specialized in anesthesia or those experienced in the care of intensive care patients. Pulmonologists, with their specific training in respiratory function management, possess crucial skills in administering deep sedation, such as that induced by propofol, as patient safety largely depends on proper airway management during the procedure.

The Complex Operative Unit of Pneumology and RICU (Respiratory Intensive Care Unit) at San Donato Hospital in Arezzo has extensive experience in the field of procedural analgesia.

This study is driven by the need to generate scientific evidence supporting effective and safe alternatives for analgosedation managed by pulmonologists during bronchoscopic procedures. The aim is to consolidate and expand upon preliminary studies in the literature, with the goal of ensuring optimal sedation even in the absence of anesthesia assistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged > 18 years;
2. Patients able to understand and sign an informed consent to participation and data collection.
3. Patients who have to undergo bronchoscopy, with or without echendoscopy, scheduled in the election, for diagnostic - staging reasons (BL or BAL with microbiological research, endobronchial biopsies, transbronchial biopsies in EBUS/EUS, EBUS/EUS-TBNA ilo-mediastinal lymph node station).
4. Patients who must undergo bronchoscopy, scheduled as an elective, for therapeutic reasons (bronchial toilet, mechanical or laser-assisted airway recanalisation)

Exclusion Criteria:

1. Patients unable to understand and sign an informed consent to participation and data collection.
2. Interventional procedures performed as a matter of urgency or without prior adequate time to clarify the methodology and objectives of the study.
3. Hypersensitivity to investigational drugs (propofol, pethidine, midazolam, local anaesthetics such as lidocaine).
4. Pre-existing haemodynamic instability or clinical conditions that may predispose to such instability during the procedure. This includes patients with acute coronary syndrome within the last 4-6 weeks, those requiring treatment with inotropes or vasoactive drugs to maintain a PAS>90 mmHg, and patients with heart failure with reduced ejection fraction (FE <40%), as defined by ESC guidelines.
5. Compromised respiratory exchanges already present before the procedure, including those requiring non-invasive ventilation (NIV), high-flow oxygen therapy via nasal cannulae (HFNC), those hospitalised for severe acute respiratory failure and patients on continuous home oxygen therapy (h24). This exclusion is necessary to avoid potential bias that could influence the study results and compromise their interpretation.
6. Inability to spontaneously protect the airways and manage bronchial secretions.
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Desaturation Index | Trough study completion, an average of 2 years
  The primary endpoint of this study is to evaluate and compare the desaturation index (SpO2 < 90% for at least 30 seconds) between the two drug regimens. The analysis will be conducted both across all procedures and stratified by type (interventional vs simple);

SECONDARY OUTCOMES:
Blood Pressure | Trough study completion, an average of 2 years
  This involves comparing the rates of peri- and post-procedural complications between the two treatment arms.
  * Hypotension defined by a systolic blood pressure <90 mmHg or a diastolic blood pressure <50 mmHg.
  * Hypotension requiring fluid therapy, vasoactive/inotropic therapy (yes or not).
Heart Rate | Trough study completion, an average of 2 years
  This involves comparing the rates of peri- and post-procedural complications between the two treatment arms.
  - Bradycardia defined as a rate <50 bpm requiring fluid therapy, vasoactive/inotropic therapy;
Respiratory Effects | Trough study completion, an average of 2 years
  This involves comparing the rates of peri- and post-procedural complications between the two treatment arms.
  - Respiratory effects: bronchospasm or wheezing requiring systemic corticosteroids, aerosolized or systemic bronchodilator therapy (e.g., beta agonists, magnesium sulphate).
Time in the recovery area | Trough study completion, an average of 2 years
  Time spent in the recovery area (in minutes)
A postanesthetic recovery score (Aldrete) | Trough study completion, an average of 2 years
  Patient recovery assessed by Aldrete score. It evaluates a patient's recovery after anesthesia based on five criteria: activity, respiration, circulation, consciousness, and oxygen saturation. Each criterion is scored from 0 to 2, resulting in a total score ranging from 0 (minimum) to 10 (maximum).
  Investigators will consider patient recovery achieved with an Aldrete score ≥9.
Rapid On Site Evaluation results | Trough study completion, an average of 2 years
  i.e.: procedure with suitable sample (Yes or Not)
Total desaturation time | Trough study completion, an average of 2 years
  Total desaturation time is defined as the cumulative time a patient's oxygen saturation (SpO2) falls below a predefined threshold (SpO2<90%) during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- San Donato Hospital, Arezzo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clarkson K, Power CK, O'Connell F, Pathmakanthan S, Burke CM. A comparative evaluation of propofol and midazolam as sedative agents in fiberoptic bronchoscopy. Chest. 1993 Oct;104(4):1029-31. doi: 10.1378/chest.104.4.1029. PMID 8404160
- [Result] Ozturk T, Cakan A, Gulerce G, Olgac G, Deren S, Ozsoz A. Sedation for fiberoptic bronchoscopy: fewer adverse cardiovascular effects with propofol than with midazolam. Anasthesiol Intensivmed Notfallmed Schmerzther. 2004 Oct;39(10):597-602. doi: 10.1055/s-2004-825919. PMID 15486802
- [Result] Clark G, Licker M, Younossian AB, Soccal PM, Frey JG, Rochat T, Diaper J, Bridevaux PO, Tschopp JM. Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. Eur Respir J. 2009 Dec;34(6):1277-83. doi: 10.1183/09031936.00142108. Epub 2009 May 14. PMID 19443532
- [Result] Lo YL, Lin TY, Fang YF, Wang TY, Chen HC, Chou CL, Chung FT, Kuo CH, Feng PH, Liu CY, Kuo HP. Feasibility of bispectral index-guided propofol infusion for flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2011;6(11):e27769. doi: 10.1371/journal.pone.0027769. Epub 2011 Nov 23. PMID 22132138
- [Result] Roelandt P, Haesaerts R, Demedts I, Bisschops R. Implementation of the Aldrete score reduces recovery time after non-anesthesiologist-administered procedural sedation in gastrointestinal endoscopy. Endosc Int Open. 2022 Dec 15;10(12):E1544-E1547. doi: 10.1055/a-1964-7458. eCollection 2022 Dec. PMID 36531676
- [Result] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Result] Allocca V, Guidelli L, Galgano A, Benedetti L, Fabbroni R, Bianco A, Paladini P, Scala R. Safety and Diagnostic Yield of Medical Pleuroscopy (MP) Performed under Balanced Analgosedation by a Pneumological Team Compared to Video-Assisted Thoracic Surgery (VATS): A Retrospective Controlled Real-Life Study (TORAPO). Diagnostics (Basel). 2024 Mar 7;14(6):569. doi: 10.3390/diagnostics14060569. PMID 38534990
- [Result] Maffucci R, Maccari U, Guidelli L, Benedetti L, Fabbroni R, Piccoli B, Bianco A, Scala R. Pulmonologist-Administered Balanced Propofol Analgosedation during Interventional Procedures: An Italian Real-Life Study on Comfort and Safety. Int J Clin Pract. 2022 Jun 13;2022:3368077. doi: 10.1155/2022/3368077. eCollection 2022. PMID 35814307
- [Result] Wang Z, Hu Z, Dai T. The comparison of propofol and midazolam for bronchoscopy: A meta-analysis of randomized controlled studies. Medicine (Baltimore). 2018 Sep;97(36):e12229. doi: 10.1097/MD.0000000000012229. PMID 30200147
- [Result] Ebert TJ. Sympathetic and hemodynamic effects of moderate and deep sedation with propofol in humans. Anesthesiology. 2005 Jul;103(1):20-4. doi: 10.1097/00000542-200507000-00007. PMID 15983452
- [Result] Fabus MS, Sleigh JW, Warnaby CE. Effect of Propofol on Heart Rate and Its Coupling to Cortical Slow Waves in Humans. Anesthesiology. 2024 Jan 1;140(1):62-72. doi: 10.1097/ALN.0000000000004795. PMID 37801625
- [Result] Lichtenbelt BJ, Mertens M, Vuyk J. Strategies to optimise propofol-opioid anaesthesia. Clin Pharmacokinet. 2004;43(9):577-93. doi: 10.2165/00003088-200443090-00002. PMID 15217302
- [Result] Williams TJ, Bowie PE. Midazolam sedation to produce complete amnesia for bronchoscopy: 2 years' experience at a district general hospital. Respir Med. 1999 May;93(5):361-5. doi: 10.1016/s0954-6111(99)90320-7. PMID 10464905
- [Result] Zomorodi K, Donner A, Somma J, Barr J, Sladen R, Ramsay J, Geller E, Shafer SL. Population pharmacokinetics of midazolam administered by target controlled infusion for sedation following coronary artery bypass grafting. Anesthesiology. 1998 Dec;89(6):1418-29. doi: 10.1097/00000542-199812000-00020. PMID 9856717
- [Result] Somma J, Donner A, Zomorodi K, Sladen R, Ramsay J, Geller E, Shafer SL. Population pharmacodynamics of midazolam administered by target controlled infusion in SICU patients after CABG surgery. Anesthesiology. 1998 Dec;89(6):1430-43. doi: 10.1097/00000542-199812000-00021. PMID 9856718
- [Result] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Result] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Result] Baughman RP, Dohn MN, Loudon RG, Frame PT. Bronchoscopy with bronchoalveolar lavage in tuberculosis and fungal infections. Chest. 1991 Jan;99(1):92-7. doi: 10.1378/chest.99.1.92. PMID 1898648
- [Result] Lachant DJ, Croft DP, McGrane Minton H, Hardy DJ, Prasad P, Kottmann RM. The clinical impact of pneumocystis and viral PCR testing on bronchoalveolar lavage in immunosuppressed patients. Respir Med. 2018 Dec;145:35-40. doi: 10.1016/j.rmed.2018.10.021. Epub 2018 Oct 22. PMID 30509714
- [Result] Postmus PE. Bronchoscopy for lung cancer. Chest. 2005 Jul;128(1):16-8. doi: 10.1378/chest.128.1.16. No abstract available. PMID 16002910